# University of Wisconsin-Madison Consent to Participate in Research (Fathers)

**Study Title for Participants:** Pathways for Parents after Incarceration Study

Formal Study Title: R00 Intervention Feasibility Study - Fatherhood after Prison: Healthy Children and

**Families** 

**Lead Researcher:** Dr. Pajarita Charles (phone: 608-263-3834; email: paja.charles@wisc.edu)

Where Lead Researcher Works: University of Wisconsin-Madison

| Participant Name | Date |
|------------------|------|

#### Invitation

We invite you and your child to be in a study about fatherhood after incarceration. The study is being done at the University of Wisconsin-Madison in partnership with JustDane, previously known as Madison-area Urban Ministry, and Anesis Therapy. We are inviting you because you 1) have been recently released from jail or prison (approximately in the last 3 years), 2) have a child (between the ages of 3 and 17), 3) play a parenting role with your child in some way, and 4) are 18 years of age or older.

The purpose of this form is to give you information needed to decide whether to be in the study. Please ask questions about anything that is unclear. You can talk to your family and friends before deciding if you want to be in the study. When we have answered all your questions, you can decide if you want to be in the study. This process is called "informed consent."

# Why are researchers doing this study?

The purpose of this study is to learn how to better support fathers and their families after incarceration. We think this can be done with reentry services that focus on parenting and problem solving. This research is being done because children with incarcerated parents often experience problems, but less is known about children with parents who have been released from prison or jail. There are not a lot of programs for children and families who have had an incarcerated parent. Learning about new options for reentry services that support the entire family may help make the parent's reentry easier on children and families. About 20 families will be in the study.

# What will happen in this study?

Pathways for Parents after Incarceration (P4P) is a community-based program that seeks to offer fathers the skills for positive father engagement and reentry success. It uses a curriculum that comes from a prison-based program, Parenting Inside Out (PIO). PIO is an evidence-based, cognitive-behavioral parent management skills training program made for incarcerated parents. It was developed by a group of scientists, policy makers, practitioners, and instructional designers. Both the information in the program and the way that information is presented come from research and practice. P4P uses eight key lessons from the original PIO curriculum that have been identified as being most helpful. They were selected by people with lived experience and by our research team. The topics focus on effective listening, speaking, and problem-solving skills, emotion regulation, and family engagement. The program will offer these 8 lessons weekly on a weekday evening for two hours. The course will be led by 1 parent coach and 1 assistant coach who will be trained to deliver the program by the PIO parent organization, The Pathfinder Network. We will also provide gift cards to compensate you for your time in the program and money to cover the cost of a meal during our time together each week.

IRB Approval Date: 9/10/2021 University of Wisconsin – Madison In addition to the classroom part of the program, each week, participants will be invited to join a peer support group led by two counselors from Anesis Therapy. This part of the program is rooted in systems therapy and uses narrative therapy, trauma focused cognitive therapy, motivational interviewing and cultural perspectives to support fathers. The groups are designed to promote people's ability to identify their values and skills so they can effectively overcome the challenges they face during reentry. The peer group sessions will be 45-60 minutes long and will take place after the 2-hour PIO class.

Both the PIO class and the peer support group will be conducted virtually through a video-call format. The parent coaches and counselors are trained in the program we are using. However, because we are using a third-party program to do this, we cannot guarantee full confidentiality. We also want to emphasize that even though we are doing remote, virtual sessions, none of it will be recorded and only those on the call with you will be able to see or hear you. In other words, we will never record any video or audio from the classes or groups.

The third and final piece of the program includes the opportunity for fathers and their families to engage in recreational, family-focused activities. P4P will provide you and your family with themed kits, such as arts, literacy, or games, or connect you with other community groups for these activities. We expect such activities to take place virtually because of the COVID-19 virus.

If you want to be in the study, we will ask you some questions about yourself and your child at the beginning of the study (before beginning the program), immediately upon graduation from the program, and 3 months later.. We will ask you questions about your relationship with your child, your feelings about spending time with your child, and your personal background. You may skip any questions in the interview that you do not want to answer. When we interview you after graduation and 3 months later, there are several questions that we will ask that we would like your permission to audio record. We will not video record you.

Also, we would like to have your permission to use exact quotes that either you or the child say. We would also like permission to get photos of you and your children. Sometimes these quotes, or the words that you say, would not be attached to your name or other identifying information. But in other cases, we would want to connect your words to the photos. Your quotes and photos might be used as part of our research and for writing reports and papers and sharing information in presentations.

As part of the project, we would like your permission about something else. We would like access to your Consolidated Court Automation Programs (CCAP) information. We can get this information using your name and birth date. CCAP is the criminal record web site for Wisconsin that anyone can access. This CCAP information will be linked to other information that we collect in this study. All of this information collected during the study will be de-identified. In other words, we will not attach names to the information. We will keep it all for future research and will not ask for permission from you, your child, or your child's caregiver to use it in the future.

Because of the study procedures and because it is funded by the National Institute of Health, the program is qualified as a clinical trial. Information from the study will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

## How long will I be in this study?

You will be part of the study for about 9 weeks and then we will follow up with you 3 months later. We will interview you today and then meet with you weekly for the P4P program. Each week day seven in gradion.

session will last for about 3 hours. In addition, it will take about 2 hours to ask you questions before the program begins, at the end of the program (after graduation), and 3 months later.

# Do I have to be in the study? What if I say "yes" now and change my mind later?

No, you do not have to be in this study. Taking part in research is voluntary and totally up to you. This means that you decide if you want to be in the study. If you decide now to be part of the study, you can choose to leave the study at any time. Let the researchers know if you want to leave the study.

If you decide not to be part of the study, or if you choose to leave the study, your choice will not affect any relationship you have with UW-Madison, JustDane, Anesis Therapy, or with any services you are receiving from the Department of Corrections. It also will not affect any relationship you have with any other organizations or any services you receive from them. We will not give any information about whether or not you participate to probation officers. Whether or not you participate is completely up to you and will have no effect on your sentence or parole. No matter what decision you make, and even if your decision changes, there will be no penalty to you. You will not get in any trouble or lose services or any legal rights.

# Will being in this study help me in any way?

Being in this study will not help you directly. Your participation in the study may help other people in the future by letting us learn more about fathers and their families after incarceration.

#### What are the risks?

There is a risk that your information could become known to someone not part of the study. If this happens, it could hurt your reputation. This could also affect your relationships with family and friends. It could affect your employment or make it harder to get insurance or a job. Also, you might become tired or frustrated because of the length of the study. To avoid that, the researcher will let you know how long we expect the activities to take during the consent process. You will be allowed to take breaks during the study activities if you want. In case you tell us about illegal behavior while you are in the study, we have a Certificate of Confidentiality to keep this information confidential. The only instance where we may need to break confidentiality is if abuse or neglect of a child is witnessed or suspected while in the home. This includes anything that is seen over the video camera. Because of how some of the questions are asked, you may tell us personal, sensitive, or identifiable information when you answer the interview questions. If you share personal information, we will store it separately from the study data. We will also make sure no one can figure out your identity in any published work.

#### Will being in this study cost me anything?

There is no cost for you to be a part of this study.

## Will I be paid or receive anything for being in this study?

You will have the potential to receive up to \$165 for participation in the study. Participants will receive \$20 at baseline data collection, \$10 for every class that they attend (up to a total of 8 classes, or \$80), \$25 for post-program data collection, and \$40 for 3-month follow-up data collection.

#### How will researchers protect my information?

We have strict rules to protect your personal information. We will limit who has access to your name, address, phone number, and other information that can identify you. We will store this information securely. We may publish and present what we learn from this study, but none of this information will identify you directly without your permission. As discussed above, we would like permission to share your photos and quotes in some cases.

Additionally, after the removal of identifiable private information, we may use the collected information for future research studies or distributed to another investigator for future research studies. If we do this, we will not obtain any additional informed consent from you or a legally authorized representative, if this might be a possibility.

However, we cannot promise total confidentiality. Federal or state laws may permit or require us to show information to university or government officials responsible for making sure this study is safe.

## Will the information I give be confidential?

Confidentiality cannot be guaranteed in a group setting or when done using a 3<sup>rd</sup> party video-call software; however, we will keep information shared during the session private. Outside of the program, the information you give will be shared only with the research team. However, the interviewer must make a report to the appropriate authorities if they have reasonable cause to believe that child abuse or neglect is occurring, as required by law. They may also need to make a report to the authorities if you threaten to hurt yourself or someone else.

To help us protect your privacy, we have a Certificate of Confidentiality from the National Institutes of Health. It covers your information from the time you start being part of this study. The researchers with this Certificate may not disclose or use information or documents that may identify you. This includes in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence. For example, if there is a court subpoena, we cannot release information unless you have given your permission for this use. This means that none of this information can be used as evidence in court. Information or documents protected by this Certificate cannot be shared with anyone else who is not part of the research. An exception is if there is a federal, state, or local law that requires disclosure (such as to report child abuse or diseases). But the information can't be used for federal, state, or local civil, criminal, administrative, legislative, or other proceedings. It is ok if you have agreed to let us share this information. Or you may want us to share information that will be used for other research, as allowed by federal regulations protecting research subjects. The Certificate of Confidentiality cannot stop us from sharing information about child abuse, or neglect or harm to yourself or other people. We are legally required by federal, state, or local laws to share this information.

## What if I have questions?

The person doing this study is Dr. Pajarita Charles. You may ask any questions you have now. If you have questions later, please feel free to call her at 608-263-3834.

If you are not satisfied with the response of the research team, have more questions, or want to talk with someone about your rights as a research participant, you should contact the Education and Social/Behavioral Science IRB Office at 608-263-2320.

## Agreement to Participate in the Research Study

If you sign the line below, it means that:

- You have read this consent form.
- You have had a chance to ask questions about the research study, and the research team has answered your questions.
- You want to be in this study.
- You give permission to have some interview questions audio recorded.
- You give permission for the researchers to use photos of you and/or your child when sharing findings from the study (INITIAL HERE):

| Printed Name of Adult Participant | |
|---|---|
| Signature of Adult Research Participant | Date |
| you sign the line below, it means that: • You have legal guardianship of the child listed by | pelow and you are able to give conse |
| child | |
| child Printed Name of Child Participant | Child Participant's Date of Birth |

\*\*You will receive a copy of this form\*\*